CLINICAL TRIAL: NCT00768261
Title: Corticolimbic Degeneration and Treatment of Dementia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01MH060883-06 (NIH)
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Results first posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Dementia
Keywords: Dementia of the Alzheimer type
MeSH Terms: conditions — Dementia | interventions — Memantine; Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Very Mild to Mild DAT Untreated (No Intervention): Group 1) subjects with very mild (CDR 0.5) to mild (CDR 1) DAT that are untreated with either cholinesterase inhibitors or memantine
- Very Mild-Mild DAT Treated W/ Donepezil (Active Comparator): Group 2) subjects with very mild (CDR 0.5) to mild (CDR 1) DAT that are treated with Donepezil (Aricept®).
  Interventions: Drug: Donepezil (Aricept®)
- Very Mild-Mild DAT Treated W/Combination (Active Comparator): Group 3) subjects with very mild (CDR 0.5) to mild (CDR 1) DAT that are treated with the combination of Donepezil (Aricept®) and Memantine (Namenda®)
  Interventions: Drug: Memantine (Namenda®); Drug: Donepezil (Aricept®)
- Nondemented Comparison Subjects (No Intervention): Group 4) nondemented comparison subjects.

INTERVENTIONS:
Drug: Memantine (Namenda®) — Drug treatment will begin with 5 mg/day of donepezil for six weeks. After six weeks of such treatment, the subjects symptoms will be re-evaluated and any side-effects of treatment assessed and recorded. If no serious side-effects of donepezil are encountered, the dose of donepezil will be increased to 10 mg/day. For subjects prescribed the combination of donepezil and memantine, memantine (20 mg/day) will be added to the drug treatment regimen after the dose of donepezil has been established (i.e., at six weeks). Again, memantine will be initially started at 10 mg/day and increased to its full dose only if no serious side-effects are encountered.
  Other Names: Namenda
  Arms: Very Mild-Mild DAT Treated W/Combination
Drug: Donepezil (Aricept®) — 5mg/day for six weeks and if no serious side-effects increased to 10mg/dy.
  Other Names: Aricept
  Arms: Very Mild-Mild DAT Treated W/ Donepezil; Very Mild-Mild DAT Treated W/Combination

SUMMARY:
The overall purpose of this research is to determine if there is a relationship between your symptoms of Dementia of the Alzheimers type and changes in the size and shape of certain brain structures during combined Donepezil (Aricept®) and Memantine (Namenda®) treatment.

DETAILED DESCRIPTION:
In this study we will be using Memantine (Namenda®) in an investigational fashion with individuals with very mild to mild dementia. Donepezil (Aricept®) is approved by the Food and Drug Administration for the treatment of Alzheimers disease. Memantine (Namenda®) is currently approved by the Food and Drug Administration for moderate and severe dementia only. This study may be instrumental in the development of a new therapy for others with similar conditions, and to determine whether Memantine (Namenda®) will be helpful to individuals with very mild to mild dementia.

Specific Aim 1. To determine what neuroanatomical measures are most strongly correlated with the progression of clinical and cognitive deficits in patients with dementia of the Alzheimer type (DAT). To accomplish this aim, we will use high-resolution magnetic resonance (MR) imaging and the tools of computational anatomy to assess changes in the structure of selected subcortical (e.g., hippocampus) and cortical (e.g., parahippocampal gyrus and cingulate gyrus) structure along with clinical and cognitive measures of dementia severity in subjects with very mild-to-mild DAT. Specific Aim 2 - To determine whether cholinesterase inhibitors and memantine can slow disease progression in DAT subjects. To accomplish this aim, we will use MR imaging and the tools of computational anatomy to compare the rate of change in the neuroanatomical measures listed above in 1) untreated DAT subjects, 2) DAT subjects treated with donepezil alone, and 3) DAT subjects treated with the combination of donepezil and memantine.

ELIGIBILITY:
Inclusion Criteria: 1) meets National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association(NINCDS-ADRDA) Alzheimer's criteria for dementia of the Alzheimer's type (DAT), 2) Clinical Dementia Rating (CDR) score of 0.5 or 1, 3) 50-80 years of age, 4) able to give informed consent or has a primary caregiver or legal guardian, who can give informed consent.

Exclusion Criteria: 1) other psychiatric (e.g., depression) or neurological (e.g., CVA) disorders that would confound the assessment of dementia symptoms, 2) history of loss of consciousness, and 3) unstable or severe medical illness (e.g., hepatotoxicity) that would make donepezil or memantine treatment or participation in other aspects of the study unsafe.

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Morris, MD, Principal Investigator — Washington University School of Medicine

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 39 subjects enrolled in Group3.14 maps have passed inspection for quality and are included in final analysis. Subject data from a previously published study of donepezil(Wang et al.,2010) with 18 very mild dementia of the Alzheimer's type patients treated with donepezil,14 untreated with mild DAT, and 56 cognitively normal individuals are included.
Groups:
- 1 Very Mild to Mild DAT Untreated: Group 1) subjects with very mild (CDR 0.5) to mild (CDR 1) DAT that are untreated with either cholinesterase inhibitors or memantine
- 2 Very Mild to Mild DAT Treated With Donepezil: Group 2) subjects with very mild (CDR 0.5) to mild (CDR 1) DAT that are treated with donepezil.
  Donepezil (Aricept®): 5mg/day for six weeks and if no serious side-effects increased to 10mg/dy.
- 3 Very Mild to Mild DAT Treated With the Combination: Group 3) subjects with very mild (CDR 0.5) to mild (CDR 1) DAT that are treated with the combination of donepezil and memantine.
  Memantine (Namenda®): Drug treatment will begin with 5 mg/day of donepezil for six weeks. After six weeks of such treatment, the subjects symptoms will be re-evaluated and any side-effects of treatment assessed and recorded. If no serious side-effects of donepezil are encountered, the dose of donepezil will be increased to 10 mg/day. For subjects prescribed the combination of donepezil and memantine, memantine (20 mg/day) will be added to the drug treatment regimen after the dose of donepezil has been established (i.e., at six weeks). Again, memantine will be initially started at 10 mg/day and increased to its full dose only if no serious side-effects are encountered.
  Memantine (Namenda®): Initial dose of 10mg/day and increased to full dose of 20mg/day if no serious side-effects
- 4 Nondemented Comparison Subjects.: Group 4) nondemented comparison subjects.
Period: Overall Study
Arm/Group | 1 Very Mild to Mild DAT Untreated | 2 Very Mild to Mild DAT Treated With Donepezil | 3 Very Mild to Mild DAT Treated With the Combination | 4 Nondemented Comparison Subjects.
Started | 14 | 18 | 39 | 56
Completed | 14 | 18 | 14 | 56
Not Completed | 0 | 0 | 25 | 0

BASELINE CHARACTERISTICS:
Population: Group 3; 39 subjects initially included. 8 subjects ineligible at initial assessment. 8 didn't have a follow-up MR scans for reasons; being deceased at the eos, refusal to scan, being unable to complete scanning due to discomfort. 5 subjects excluded due to poor baseline MR quality. 4 more scans excluded due to poor longitudinal mapping quality
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Very Mild to Mild DAT Untreated | 2 Very Mild to Mild DAT Treated With Donepezil | 3 Very Mild to Mild DAT Treated With the Combination | 4 Nondemented Comparison Subjects. | Total
Number analyzed (Participants) | 14 | 18 | 14 | 56 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 0 | 0 | 2
  >=65 years | 13 | 17 | 14 | 56 | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 6 | 35 | 55
  Male | 8 | 10 | 8 | 21 | 47
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 18 | 14 | 56 | 102

OUTCOME MEASURES:

1. Primary Outcome: Rate of Change of Hippocampal Volume Slope
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: mm^3/year
Arm/Group | 1 Very Mild to Mild DAT Untreated | 2 Very Mild to Mild DAT Treated With Donepezil | 3 Very Mild to Mild DAT Treated With the Combination | 4 Nondemented Comparison Subjects.
Number analyzed (Participants) | 14 | 18 | 14 | 56
mm^3/year
  left hippocampal volume slope | -70.2418748 (31.4801034) | -88.4738591 (52.2621175) | -94.0768115 (48.349487) | -46.9484805 (83.5825530)
  right hippocampal volume slope | -99.9437062 (65.1619838) | -94.3258652 (44.7959659) | -125.0687876 (72.5509442) | -80.0840066 (130.3453711)
Statistical Analysis 1: Comparison: 1 Very Mild to Mild DAT Untreated vs 2 Very Mild to Mild DAT Treated With Donepezil vs 3 Very Mild to Mild DAT Treated With the Combination vs 4 Nondemented Comparison Subjects; Test type: Other; p = 0.095, ANOVA; df= 3,92

2. Secondary Outcome: Comparison of Combined DAT Patients' Mean (SD) Hippocampal Volume Slope (mm^3/Year) Rate of Change
Description: The ADAS-Cog evaluates cognition and differentiates normal from impaired cognitive functioning. The total score is the summed number of errors in each task. The greater the impairment, the greater the score. We combined the dementia of the Alzheimer's type patients receiving all treatments together and grouped them into 3 subgroups according to the rates of change(roc) of their ADAS-Cog scores. To determine trends in hippocampal volume atrophy over time we compared the patients showing most negative ADAS-Cog rate of change (improving), patients with most positive ADAS-cog roc (worsening), patients with intermediate, near-zero ADAS-Cog roc (stable) .
Time Frame: two years
Population: We combined the DAT patients who received any treatment (donepezil or combined) & used the annual roc in ADAS-Cog to equally separate them into 3 subgroups; improving (1/3 negative ADAS-Cog roc), stable (1/3 near-zero ADAS-Cog change) & worsening (1/3 positive ADAS-Cog change).
Measure: Mean (Standard Deviation); unit: (mm^3/year)
Groups:
- Improved; Worsening; Stable: Response group by ADAS-Cog rates
Arm/Group | Improved | Worsening | Stable
Number analyzed (Participants) | 10 | 11 | 11
(mm^3/year)
  left hippocampal volume slope | -70 (56) | -106 (55) | -100 (37)
  right hippocampal volume slope | -77 (51) | -141 (78) | -105 (34)
Statistical Analysis 1: Comparison: Improved vs Stable; There would be a treatment effect on the changes of hippocampal measures over time. Repeated measures ANOVA on hippocampal volume slopes with hemisphere as a within-subject repeated factor, and treatment group as the main effect; Test type: Other; p = 0.066, ANOVA
Statistical Analysis 2: Comparison: Improved vs Worsening; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.009, ANOVA
Statistical Analysis 3: Comparison: Worsening vs Stable; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.30, ANOVA
Statistical Analysis 4: Comparison: Improved vs Worsening vs Stable; RM-ANOVA on hippocampal volume slope; Test type: Other; p = 0.0288, Repeated Measures ANOVA

ADVERSE EVENTS:
Arm/Group | 1 Very Mild to Mild DAT Untreated | 2 Very Mild to Mild DAT Treated With Donepezil | 3 Very Mild to Mild DAT Treated With the Combination | 4 Nondemented Comparison Subjects.
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/18 | 0/14 | 0/56
Other Adverse Events (participants affected / at risk) | 0/14 | 0/18 | 0/14 | 0/56

LIMITATIONS AND CAVEATS:
Interpretation of results limited to evaluating overall effects in naturalistic groups undergoing 2 drug treatments;Insufficient subjects to determine possible existence of DAT patient subgroups showing drug-specific slowing of disease progression

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-08-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT00768261/Prot_SAP_000.pdf